CLINICAL TRIAL: NCT04241471
Title: Incision and Loop Drainage Utilizing a Novel Technique for Management of Cutaneous Abscess in an Adult Population: a Randomized Control Trial
Brief Title: Incision and Loop Drainage Utilizing a Novel Technique for Management of Cutaneous Abscess in an Adult Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study published rendering this protocol/study obsolete.
Sponsor: bryan malcolm (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, bryan malcolm, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20200046H
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Abscess; Drain Abscess
Keywords: Emergency Medicine; Abscess; Incision and Drainage; Incision and Loop Drainage; Sterile Glove
MeSH Terms: conditions — Abscess; Surgical Wound | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- traditional incision and drainage (I&D) (Active Comparator)
  Interventions: Device: traditional incision and drainage (I&D)
- incision and loop drainage (Experimental): incision and loop drainage utilizing the rolled ring of a sterile glove technique
  Interventions: Procedure: incision and loop drainage

INTERVENTIONS:
Procedure: incision and loop drainage — incision and loop drainage utilizing the rolled ring of a sterile glove technique
  Arms: incision and loop drainage
Device: traditional incision and drainage (I&D) — traditional incision and drainage (I&D)
  Arms: traditional incision and drainage (I&D)

SUMMARY:
When using the rolled ring of a sterile glove as a loop drain in incision and loop drainage, is it superior to incision and drainage for treatment of a cutaneous abscess in 18 to 65 year-old patients presenting to the Emergency Department, Family Health Clinic, Family Medicine Residency Clinic, or Internal Medicine Clinic?

Hypothesis: When treating a cutaneous abscess, incision and loop drainage utilizing the rolled ring of a sterile glove as a loop drain is superior to the standard (incision and drainage) yielding a treatment failure rate of 1% at seven to ten days.

DETAILED DESCRIPTION:
Practicing medicine in an austere environment is fraught with challenges. One primary challenge is that clinicians will frequently be practicing without the supplies needed for specific indicated purpose. For treatment of a cutaneous abscess, sterile gloves are readily available whether at home or when deployed. It can be much more difficult to come across a penrose or vessel loop. In addition, follow up for wound repacking and reassessment is a struggle. Patients may have to move from location to location or have work hours that make it difficult to return to the clinic. The loop technique utilizing the rolled ring of a sterile glove solves both of these problems. Sterile gloves are always available and the Loop technique requires little to no follow up. Additional benefits include: subjects may experience less pain, improved cosmesis, faster healing, and decreased complication rates with incision and loop drainage utilizing the rolled ring of a sterile glove compared to traditional incision and drainage.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active Duty and DoD beneficiaries aged 18 to 65 years old.
* Abscess that requires drainage.

Exclusion Criteria:

* Abscess of the hand, foot, or face, immunocompromised by disease or medications.
* Temperature greater than 100.4 degrees Fahrenheit.
* Systolic blood pressure less than 90 mmHG.
* Abscess is too small to treat with incision and drainage (as seen on ultrasound).
* Patient is too ill to be included in the study determined by clinical judgement of the treating provider.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Treatment effectiveness | 30 days post-procedure
  A record review will be performed to identify patients that had to return to the Emergency Department up to 30 days after the procedure due to complications. Attempts will be made to contact patients who fail to follow up. If unable to contact, a record review will be conducted in attempt to ascertain abscess status. If these measures are unsuccessful, patient treatment will be considered a success.
  Record Review: Treatment failure will be defined as need for repeat drainage, intravenous antibiotic, hospitalization or surgical treatment within 7 days.
Subject pain: Visual Analogue Scale | Pre-procedure, mid-procedure, post-procedure
  Data will be collected using the VAS. Patients mark will be measured in millimeters and recorded.
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Lower scores mean a better outcome and higher scores mean greater pain severity.
Provider satisfaction: Visual Analogue Scale | post-procedure
  Data will be collected using the VAS. Provider mark will be measured in millimeters and recorded.
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. In this case, higher scores mean a better outcome (satisfaction) and lower scores mean less satisfaction.
Subject satisfaction: Visual Analogue Scale | 7-10 day follow-up
  Data will be collected using the VAS. Subject mark will be measured in millimeters and recorded.
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. In this case, higher scores mean a better outcome (satisfaction) and lower scores mean less satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Study Director — United States Air Force

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] Aprahamian CJ, Nashad HH, DiSomma NM, Elger BM, Esparaz JR, McMorrow TJ, Shadid AM, Kao AM, Holterman MJ, Kanard RC, Pearl RH. Treatment of subcutaneous abscesses in children with incision and loop drainage: A simplified method of care. J Pediatr Surg. 2017 Sep;52(9):1438-1441. doi: 10.1016/j.jpedsurg.2016.12.018. Epub 2016 Dec 30. PMID 28069270
- [Background] Brody AM, Gallien J, Murphy D, Marogil J. A Novel Silicon Device for the Packing of Cutaneous Abscesses. J Emerg Med. 2019 Mar;56(3):298-300. doi: 10.1016/j.jemermed.2018.12.009. Epub 2019 Jan 17. PMID 30661820
- [Background] Gottlieb M, Peksa GD. Comparison of the loop technique with incision and drainage for soft tissue abscesses: A systematic review and meta-analysis. Am J Emerg Med. 2018 Jan;36(1):128-133. doi: 10.1016/j.ajem.2017.09.007. Epub 2017 Sep 10. PMID 28917436
- [Background] Ladde JG, Baker S, Rodgers CN, Papa L. The LOOP technique: a novel incision and drainage technique in the treatment of skin abscesses in a pediatric ED. Am J Emerg Med. 2015 Feb;33(2):271-6. doi: 10.1016/j.ajem.2014.10.014. Epub 2014 Oct 16. PMID 25435407
- [Background] Leinwand M, Downing M, Slater D, Beck M, Burton K, Moyer D. Incision and drainage of subcutaneous abscesses without the use of packing. J Pediatr Surg. 2013 Sep;48(9):1962-5. doi: 10.1016/j.jpedsurg.2013.01.027. PMID 24074675
- [Background] Long B, April MD. Is Loop Drainage Technique More Effective for Treatment of Soft Tissue Abscess Compared With Conventional Incision and Drainage? Ann Emerg Med. 2019 Jan;73(1):19-21. doi: 10.1016/j.annemergmed.2018.02.006. Epub 2018 Mar 9. No abstract available. PMID 29530657
- [Background] McNamara WF, Hartin CW Jr, Escobar MA, Yamout SZ, Lau ST, Lee YH. An alternative to open incision and drainage for community-acquired soft tissue abscesses in children. J Pediatr Surg. 2011 Mar;46(3):502-6. doi: 10.1016/j.jpedsurg.2010.08.019. PMID 21376200
- [Background] Ozturan IU, Dogan NO, Karakayali O, Ozbek AE, Yilmaz S, Pekdemir M, Suner S. Comparison of loop and primary incision & drainage techniques in adult patients with cutaneous abscess: A preliminary, randomized clinical trial. Am J Emerg Med. 2017 Jun;35(6):830-834. doi: 10.1016/j.ajem.2017.01.036. Epub 2017 Jan 22. PMID 28162873
- [Background] Schechter-Perkins EM, Dwyer KH, Amin A, Tyler MD, Liu J, Nelson KP, Mitchell PM. Loop Drainage Is Noninferior to Traditional Incision and Drainage of Cutaneous Abscesses in the Emergency Department. Acad Emerg Med. 2020 Nov;27(11):1150-1157. doi: 10.1111/acem.13981. Epub 2020 May 14. PMID 32406569
- [Background] Thompson DO. Loop drainage of cutaneous abscesses using a modified sterile glove: a promising technique. J Emerg Med. 2014 Aug;47(2):188-91. doi: 10.1016/j.jemermed.2014.04.035. Epub 2014 Jun 11. PMID 24928539
- [Background] Tsoraides SS, Pearl RH, Stanfill AB, Wallace LJ, Vegunta RK. Incision and loop drainage: a minimally invasive technique for subcutaneous abscess management in children. J Pediatr Surg. 2010 Mar;45(3):606-9. doi: 10.1016/j.jpedsurg.2009.06.013. PMID 20223328
- [Background] Gaspari RJ, Sanseverino A, Gleeson T. Abscess Incision and Drainage With or Without Ultrasonography: A Randomized Controlled Trial. Ann Emerg Med. 2019 Jan;73(1):1-7. doi: 10.1016/j.annemergmed.2018.05.014. Epub 2018 Aug 17. PMID 30126754
- See also: loop drainage — https://baylor.primo.exlibrisgroup.com/discovery/fulldisplay?docid=wos000445699100183&context=PC&vid=01BUL_INST:BAYLOR&lang=en&search_scope=MyInst_and_CI&adaptor=Primo%20Central&tab=Everything&query=any,contains,incision%20and%20loop%20drainage&offset=0.